CLINICAL TRIAL: NCT07233291
Title: Evaluation of Efficacy and Safety of Oral Roflumilast in Treatment of Moderate to Severe Psoriasis: a Pilot Study
Brief Title: A Pilot Study to Assess How Safe and Effective Oral Roflumilast is for Treating Moderate to Severe Psoriasis in Adults
Acronym: PSOROFLU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ahmed Ibrahim (Other)
Collaborators: Mansoura University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ahmed Ibrahim, Assistant lecturer of dermatology, Andrology, & STDs , Suez University., Mansoura University Hospital
Organization: Mansoura University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.25.06.3223.R1
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis (PsO)
Keywords: Psoriasis; Moderate to severe Psoriasis; Roflumilast; Oral Roflumilast; PDE4 Inhibitor; Plaque Psoriasis; Pilot Study; Adults
MeSH Terms: conditions — Psoriasis | interventions — Roflumilast; Tablets

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label pilot study in which all participants, both male and female, receive oral roflumilast. Participants will not be randomized to different treatments. Male and female participants will be analyzed as subgroups to explore potential sex-based differences in safety and efficacy. No placebo or comparator group is included.
Masking Description: This is an open-label study: neither the participants nor the investigators are blinded. All participants receive oral roflumilast, and both participants and study staff are aware of the treatment assignment. No placebo or comparator is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral Roflumilast for Adults with Moderate-to-Severe Psoriasis (Experimental): All participants, both male and female, will receive oral roflumilast.
  No placebo or comparator is included.
  Male and female participants will be analyzed as subgroups for exploratory safety and efficacy outcomes.
  Interventions: Drug: Oral roflumilast

INTERVENTIONS:
Drug: Oral roflumilast — Dosage: Participants will receive oral roflumilast. The initial dose is 250 mcg once daily for the first 10 days, followed by a dose escalation to 500 mcg once daily for the remainder of the 12-week treatment period.
  Route: Oral
  Schedule: Daily for 12 weeks
  Duration: 12 weeks
  Other Names: Roflumilast (generic name); Daxas (brand name in some countries); Roflumilast 500 mcg tablet (formulation identifier)

SUMMARY:
This is a 12-week, single-arm, open-label pilot study to assess the safety and preliminary efficacy of oral roflumilast in adults with moderate-to-severe plaque psoriasis. All participants, both male and female, will receive oral roflumilast starting at 250 mcg once daily for 10 days, followed by 500 mcg once daily for the remainder of the study. The primary outcome is the mean change in Psoriasis Area and Severity Index (PASI) score from baseline to Week 12. Secondary outcomes include change in body mass index (BMI) and safety assessments, including treatment-emergent adverse events, serious adverse events, and laboratory abnormalities. Male and female participants will be analyzed as subgroups.

DETAILED DESCRIPTION:
This pilot study is designed to evaluate the safety and preliminary efficacy of oral roflumilast in adults with moderate-to-severe plaque psoriasis. The study was approved by the Mansoura University Faculty of Medicine Institutional Review Board (IRB), Approval Code: R.25.06.3223.R1, and participants will be enrolled only after obtaining informed consent.

Each participant will undergo a detailed history and clinical examination, including:

Personal history: name, age, sex, occupation, residence, marital status, number of children, and special habits of medical importance.

History of present illness: onset, course, duration of psoriasis, and precipitating factors.

Medication history: nature, route, dose, compliance, duration, effect, and side effects.

Family history: psoriasis or other dermatoses.

Past medical history: associated systemic, other dermatological diseases, or major surgical operations.

Menstrual and obstetric history (for female participants).

A general clinical examination will be performed to assess overall health and exclude any systemic diseases.

The study will monitor clinical response using the Psoriasis Area and Severity Index (PASI) and record body mass index (BMI) changes. Safety will be assessed through monitoring of treatment-emergent adverse events, serious adverse events, and routine laboratory tests. Participants will attend scheduled visits throughout the 12-week treatment period, and data will be analyzed overall and by sex-based subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic patients ≥ 18 years in whom systemic therapy is indicated.
* Chronic stable plaque psoriasis.
* Patients who don't use other systemic therapy for psoriasis in the last 2 months (or naïve who didn't use any systemic therapy before).
* Safe contraception during the study.

Exclusion Criteria:

* Pregnant or lactating women, as well as women of childbearing potential not using an effective method of contraception.
* Age <18 years.
* Other concomitant psoriasis systemic treatments such as Acitretin and biologics.
* Previous systemic treatment of psoriasis in the last 2 months.
* Patients receiving inducers or inhibitors of cytochromes CYP3A4 and CYP1A.
* Other systemic diseases other than COPD, especially hepatic impairment.
* Hypersensitivity to the active substance of roflumilast or to any of its excipients
* The use of contraception with gestodene and ethinylestradiol
* Unreliable patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean change in Psoriasis Area and Severity Index (PASI) score | Baseline to Week 12
  The mean difference in PASI score from baseline to Week 12 among adults with moderate-to-severe plaque psoriasis receiving oral roflumilast. PASI is a validated composite measure of psoriasis severity assessing erythema, induration, desquamation, and affected body surface area.

SECONDARY OUTCOMES:
Change in body mass index (BMI) | Baseline to Week 12
  Mean change in BMI (kg/m²), calculated from measured weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Mohamed Elkholy, MD Dermatology, Study Chair — Faculity of Medicine, Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt